CLINICAL TRIAL: NCT03937492
Title: EFFECTIVENESS OF GRADED MOTOR IMAGERY TO PREVENT CRPS IN PATIENTS WITH DISTAL RADIUS FRACTURE AFTER SURGERY: A RANDOMIZED CONTROLLED TRIAL
Brief Title: EFFECTIVENESS OF GRADED MOTOR IMAGERY TO PREVENT CRPS IN PATIENTS WITH DISTAL RADIUS FRACTURE AFTER SURGERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ergoterapia Manoegomito Sagl (Other)
Responsible Party: Principal Investigator, Pagella Susanna, Principal Investigator, Ergoterapia Manoegomito Sagl
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Ergoterapia manoegomito
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Wrist Fracture; CRPS (Complex Regional Pain Syndromes); Distal Radius Fracture; Surgery
Keywords: GMI; CRPS; Distal radius fracture
MeSH Terms: conditions — Wrist Fractures; Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): In this group patients follow standard treatment after radius fracture plus GMI procol
  Interventions: Other: GMI protocol; Other: Standard Rehabilitation Protocol
- B group (Active Comparator): In this group patients follow standard treatment after radius fracture
  Interventions: Other: Standard Rehabilitation Protocol

INTERVENTIONS:
Other: GMI protocol — This group follow GMI program split in 3 step:
  1. left/right descrimination
  2. visual motor imagery
  3. mirror therapy
  Patients perform this exercises 3 times every day and they have checks in therapy al least twice a week.
  Arms: A group
Other: Standard Rehabilitation Protocol — This group follow standard rehabilitation protocol, with active and passive motion of upper limb structure, including hand, wrist, elbow, shoulder.
  Patients perform this exercises 3 times every day and they have checks in therapy al least twice a week.

SUMMARY:
The study would like show that patients who follow a protocol with GMI are less probability to develop CRPS

DETAILED DESCRIPTION:
Distal radius fractures (DRF) has a high frequency in adults. Studies show that the upper limb is frequently affected by CRPS, especially if is preceded by a fracture.

Recent studies suggest that changes in cortical structures can contribute to the onset of CRPS.

GMI is a approved and efficacy method in CRPS rehabilitation, because it trains modified cortical areas throught 3 stadies: left-right discrimination, visual motor imagery and mirror therapy.

Literature shows that there are any studies about GMI efficacy on prevention CRPS in DRF after surgery.

This study would like to demostrate that, appling GMI in the early stages of rehabilitation plus standard rehabilitation protocol of DRF after surgery, CRPS cases are reducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fracture after surgery
* 18 to 75 years old
* Male and female

Exclusion Criteria:

* uncompliants patients
* patients with neurological disorders or cognitive impairment
* patients with TFCC injury or both ulna and radius fractures
* patients with visually impairment
* patients who don't speak or understand oral and written italian language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-02 (Estimated); Primary Completion 2020-05-02 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Range Of Motion | Baseline and 8 weeks
  Change in active and passive range of motion about hand and wrist

SECONDARY OUTCOMES:
Patient-rated wrist/hand evaluation (prwhe) | Baseline and 8 weeks
  Decrease in difficulty of doing activities of daily living and decrease pain
Jamar hand dynamometer | Baseline and 8 weeks
  Improve strength
McGill pain questionnaire | Baseline and 8 weeks
  Decrease pain

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Pagella, Principal Investigator — Ergoterapia Manoegomito Sagl

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR